CLINICAL TRIAL: NCT00388609
Title: A Randomized, Double-blind, Placebo-Controlled, Parallel Arm, Multiple-Dose Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of BMS-646256 in Obese and High Risk Overweight Subjects
Brief Title: Multiple-dose Study to Evaluate the Efficacy, Safety and Pharmacokinetics of BMS-646256 in Obese Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB109-007
Record Dates: First submitted 2006-10-05; First posted 2006-10-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2009-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- T (Experimental): 5 mg (ST) to 50 mg (LT)
  Interventions: Drug: BMS-646256
- U (Experimental): 10 mg (ST) to 50 mg (LT)
  Interventions: Drug: BMS-646256
- V (Experimental): 25 mg (ST) to 50 mg (LT)
  Interventions: Drug: BMS-646256
- W (Experimental): 50 mg (ST and LT)
  Interventions: Drug: BMS-646256
- X (Experimental): 25 mg/d (X1 wk), 5 mg/d (X11 wks) (ST) to 50 mg (LT)
  Interventions: Drug: BMS-646256
- Z (Experimental): Open label: 50 mg/d (X 4 wks) 100 mg/wk (X8 wks) (ST) to 50 mg (LT)
  Once daily (x 4 weeks), once daily (x 8 weeks)
  Interventions: Drug: BMS-646256
- Y (Placebo Comparator): 0 mg (ST and LT)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-646256 — Tablet, Oral, Once Daily, 12 weeks treatment followed by 20 week washout (ST); up to 190 weeks treatment (LT)
  Arms: T; U; V; W; X; Z
Drug: Placebo — Tablet, Oral, Once daily, 12 weeks treatment followed by 20 week washout (ST); up to 190 weeks treatment (LT)
  Arms: Y

SUMMARY:
The purpose of this study is to learn if BMS-646256 can cause weight loss in men and women who are:

* overweight with high blood pressure or high cholesterol or
* obese

The safety of this treatment will also be studied

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages ≥18 to ≤70 years old with a Body Mass Index (BMI) ≥30 to ≤45 kg/m² OR BMI >27 to <30 kg/m² with hypertension and/or dyslipidemia defined as:
* Hypertension defined as treatment with an antihypertensive agent or mean systolic blood pressure ≥140 and ≤160 mmHg and/or diastolic blood pressure ≥ 90 and ≤ 105 mmHg
* Dyslipidemia defined as stable dose treatment with a statin, fibrate or ezetimibe for ≥ 6 weeks and/or triglycerides ≥ 150 and ≤ 600 mg/dL, LDL ≥ 130 and ≤ 300 mg/dL, or HDL < 40 mg/dL

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* history of MI in the prior 6 months
* history of heart failure
* history of symptomatic arrhythmia
* active hepatic disease
* any documented muscle disease
* history of neurological symptoms or disease (including but not limited to tremor, ataxia, dizziness, neuropathy, or episodes of confusion, history of seizures, stroke or TIA)
* known history of major psychiatric conditions (e.g. schizophrenia anxiety disorder, dementia or bipolar disorder as defined by DSM IV criteria)
* history of depression or suicide attempt or ideation
* previous history of surgical procedures for weight loss (e.g., stomach stapling, bypass)
* uncontrolled blood pressure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from the start of the study | Average of Week 11 and 12

SECONDARY OUTCOMES:
Change in body weight | Average of Week 11 and 12
BMI | Change from baseline to Week 12, Week 32, and Week 44
waist circumference | Change from baseline to Week 12, Week 32, and Week 44
hormonal measures of insulin sensitivity and safety | Percent change from baseline to Week 12, Week 32, and Week 44
blood pressure | Change from baseline to Week 12, Week 32, and Week 44
blood lipids | Change from baseline to Week 12, Week 32, and Week 44
incidence of adverse events and lab abnormalities | throughout the study
Change and percent change in body weight | at Week 32 from baseline and Week 12
Time-matched change from baseline in QTc | at Week 12 and Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (10):
  - Ucla Center For Human Nutrition, Los Angeles, California
  - Domenica M. Rubino, Md, Washington D.C., District of Columbia
  - Csra Partners In Health, Inc, Augusta, Georgia
  - Springfield Diabetes And Endocrine Center, Springfield, Illinois
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - The Center For Nutrition & Preventive Medicine, Pllc, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - Hampton Roads Center For Clinical Research Inc., Norfolk, Virginia
  - National Clinical Research, Inc., Richmond, Virginia